CLINICAL TRIAL: NCT05762198
Title: A Randomized Controlled Trial Comparing Water Vapour Thermal Therapy (Rezūm) and TURP in Men With Benign Prostatic Hyperplasia in Refractory Urinary Retention
Brief Title: Comparing Water Vapour Thermal Therapy (Rezūm) and TURP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2022.537-T
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rezūm (Active Comparator)
  Interventions: Device: Rezūm
- TURP (Active Comparator)
  Interventions: Device: TURP

INTERVENTIONS:
Device: Rezūm — In the REZUM arm, water vapour treatment is performed for all subjects under local anaesthesia.
  Arms: Rezūm
Device: TURP — In the TURP arm, all men will receive TURP operation under general or spinal anaesthesia
  Arms: TURP

SUMMARY:
This is a randomized controlled trial using a non-inferiority design with the subjects randomized 1:1 to either water vapour thermal treatment (REZUM) arm or transurethral resection of prostate (TURP) arm.

ELIGIBILITY:
Inclusion Criteria:

* Men 50-80 years
* Refractory urinary retention related to benign prostatic hyperplasia (BPH)
* On urethral Foley's catheter before treatment
* Prostate size 30-80ml on ultrasound

Exclusion Criteria:

* Prior prostate operation
* Past or current history of prostate cancer
* Strong suspicion of prostate cancer (e.g. Elevated PSA before urinary retention or abnormal prostate on DRE without workup for prostate cancer)
* Known Urethral stricture / Bladder stone / Hypocontractile bladder
* Known neurological diseases which may affect bladder function (e.g. Parkinsonism, stroke)
* Contraindicated to undergo TURP or REZUM (e.g. not fit for GA/SA, active urinary tract infection, fail to be placed in lithotomy position, uncorrectable coagulopathy, antiplatelet or anticoagulant which cannot be stopped)

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 108 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in International Prostate Symptom Score (IPSS) at 12 months after treatment | Baseline, 3 months, 6 months and 12 months after intervention
  IPSS score ranging from 0-35 (the higher the worse)

SECONDARY OUTCOMES:
Successful trial without catheter (TWOC) within 3 months | At 3 months
  Percentage of patients successfully TWOC
Complication rate | 30 days after intervention
  Assessed by Clavien-Dindo classification
Post-op quality of life score | Baseline, 3 months, 6 months and 12 months after intervention
  Change in quality of life assessed by change in International Prostate QOL score (ranges from 0 to 6, the higher the worse)
Change in voiding function in uroflowmetry | Baseline, 3 months, 6 months and 12 months after intervention
  It is assessed by maximum flow rate and post void volume in uroflowmetry
Post-op International Index of Erectile function score | Baseline, 3 months, 6 months and 12 months after intervention
  Score 1-5 (the lower the worse)
Hospital stays of procedure | On Discharge
  Measure the hours of in-patient hospitalisation
Unplanned readmission rate after operation in 30 days | 30 days after intervention
  Percentage of patients with unplanned readmission

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fung CHIU, FRCS, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng CF, Yee CH, Chan CK, Wong HM, Chiu PK, Tsu JH, Teoh JY, Ho KL. Bipolar transurethral vapourisation versus monopolar transurethral resection of prostate: a randomised controlled trial. Hong Kong Med J. 2017 Jun;23 Suppl 2(3):32-34. No abstract available. PMID 29938669
- [Background] Yee CH, Wong JH, Chiu PK, Teoh JY, Chan CK, Chan ES, Hou SM, Ng CF. Secondary hemorrhage after bipolar transurethral resection and vaporization of prostate. Urol Ann. 2016 Oct-Dec;8(4):458-463. doi: 10.4103/0974-7796.192110. PMID 28057992
- [Background] Yee CH, Wong JH, Chiu PK, Chan CK, Lee WM, Tsu JH, Teoh JY, Ng CF. Short-stay transurethral prostate surgery: A randomized controlled trial comparing transurethral resection in saline bipolar transurethral vaporization of the prostate with monopolar transurethral resection. Asian J Endosc Surg. 2015 Aug;8(3):316-22. doi: 10.1111/ases.12197. Epub 2015 Jun 3. PMID 26042336
- [Background] Yip SK, Chan NH, Chiu P, Lee KW, Ng CF. A randomized controlled trial comparing the efficacy of hybrid bipolar transurethral vaporization and resection of the prostate with bipolar transurethral resection of the prostate. J Endourol. 2011 Dec;25(12):1889-94. doi: 10.1089/end.2011.0269. Epub 2011 Sep 16. PMID 21923418
- [Background] Teo JS, Lee YM, Ho HSS. An update on transurethral surgery for benign prostatic obstruction. Asian J Urol. 2017 Jul;4(3):195-198. doi: 10.1016/j.ajur.2017.06.006. Epub 2017 Jun 15. PMID 29264231
- [Background] McVary KT, Gange SN, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Rousseau M, Beahrs JR, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Larson TR, Dixon CM, Roehrborn CG. Minimally Invasive Prostate Convective Water Vapor Energy Ablation: A Multicenter, Randomized, Controlled Study for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2016 May;195(5):1529-1538. doi: 10.1016/j.juro.2015.10.181. Epub 2015 Nov 22. PMID 26614889
- [Background] Cantrill CH, Zorn KC, Elterman DS, Gonzalez RR. The Rezum system - a minimally invasive water vapor thermal therapy for obstructive benign prostatic hyperplasia. Can J Urol. 2019 Jun;26(3):9787-9793. PMID 31180311
- [Background] McVary KT, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Pliskin M, Beahrs JR, Prall D, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Tadros NN, Gange SN, Roehrborn CG. Final 5-Year Outcomes of the Multicenter Randomized Sham-Controlled Trial of a Water Vapor Thermal Therapy for Treatment of Moderate to Severe Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2021 Sep;206(3):715-724. doi: 10.1097/JU.0000000000001778. Epub 2021 Apr 19. PMID 33872051
- [Background] McVary KT, El-Arabi A, Roehrborn C. Preservation of Sexual Function 5 Years After Water Vapor Thermal Therapy for Benign Prostatic Hyperplasia. Sex Med. 2021 Dec;9(6):100454. doi: 10.1016/j.esxm.2021.100454. Epub 2021 Oct 30. PMID 34731779
- [Background] McVary KT, Holland B, Beahrs JR. Water vapor thermal therapy to alleviate catheter-dependent urinary retention secondary to benign prostatic hyperplasia. Prostate Cancer Prostatic Dis. 2020 Jun;23(2):303-308. doi: 10.1038/s41391-019-0187-5. Epub 2019 Nov 18. PMID 31740738
- [Background] Barry MJ, Williford WO, Chang Y, Machi M, Jones KM, Walker-Corkery E, Lepor H. Benign prostatic hyperplasia specific health status measures in clinical research: how much change in the American Urological Association symptom index and the benign prostatic hyperplasia impact index is perceptible to patients? J Urol. 1995 Nov;154(5):1770-4. doi: 10.1016/s0022-5347(01)66780-6. PMID 7563343
- [Background] Ray AF, Powell J, Speakman MJ, Longford NT, DasGupta R, Bryant T, Modi S, Dyer J, Harris M, Carolan-Rees G, Hacking N. Efficacy and safety of prostate artery embolization for benign prostatic hyperplasia: an observational study and propensity-matched comparison with transurethral resection of the prostate (the UK-ROPE study). BJU Int. 2018 Aug;122(2):270-282. doi: 10.1111/bju.14249. Epub 2018 May 6. PMID 29645352
- [Background] Yu SCH, Cho C, Hung E, Wang D, Chiu P, Yee CH, Ng A. Case-Control Study of Intra-arterial Verapamil for Intraprostatic Anastomoses to Extraprostatic Arteries in Prostatic Artery Embolization for Benign Prostatic Hypertrophy. J Vasc Interv Radiol. 2017 Aug;28(8):1167-1176. doi: 10.1016/j.jvir.2017.04.004. Epub 2017 May 13. PMID 28506701